CLINICAL TRIAL: NCT05272995
Title: Recalled International Index of Erectile Function-5 Collected 3 Months Postoperatively in Assessing Preoperative Erectile Function in Patients Undergoing Radical Prostatectomy
Brief Title: Recalled International Index of Erectile Function-5 Collected Post Prostatectomy in Assessing Preop Erectile Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Stavros Kontogiannis, Consultant of Urology, University Hospital of Patras
Other Study IDs: 114/21-02-2022
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy
Keywords: Erectile dysfunction; Prostate cancer; IIEF-5; Radical prostatectomy
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IIEF-5 — The participants will be asked to complete a validated IIEF-5 questionnaire, an abridged version of the IIEF. The IIEF is a validated, brief and reliable self-administered questionnaire for assessing erectile function. Moreover, this tool is easily administered in clinical setting and demonstrates adequate sensitivity and specificity for detecting treatment-related changes in erectile function in patients with erectile dysfunction (ED).According to Rosen et al the abridged five-item version of the 15-item IIEF possesses favorable properties for detecting the presence and severity of ED for the preceding 6 months. The IIEF-5 consists of five questions, each of which is scored on a five-point ordinal scale and ED may be classified into five categories based on the calculated scores.

SUMMARY:
The accurate assessment of erectile function before radical prostatectomy, using validated questionnaires like IIEF-5, is crucial to evaluate postoperative changes in erectile function, as the preoperative erectile function is a prognostic factor for the postoperative recovery of erectile function. In clinical practice, patients usually present at the urologist's office 3 months after the operation without a preoperative IIEF-5 score and at that time the doctors ask them about their preoperative erectile function. With this study, the investigators would like to evaluate the agreement between a real-time preoperative IIEF-5 and a recalled one 3 months after radical prostatectomy.

DETAILED DESCRIPTION:
Radical prostatectomy (RP) is a widely performed procedure for patients with clinically localized prostate cancer and its most common side effects include urinary incontinence and erectile dysfunction. These two side-effects become progressively more important to health-related quality of life (HRQOL) and thus the balance between cancer control and preservation of HRQOL is challenging. The postoperative changes in erectile function are directly related with the preoperative erectile function status of the patient. The most accurate evaluation of the pretreatment erectile function is the International Index of Erectile Function-5 questionnaire. The fact that in some cases the preoperative questionnaire results are negatively affected by several factors, indicates the necessity of the assessment of the degree of agreement between real time IIEF-5 scores and retrospective IIEF-5 scores after radical prostatectomy. Frequently the andrologists do not have a preoperative IIEF-5 score in their hands and this might happen for various reasons. The main reason is that urologists ask about the preoperative erectile function often with just a simple question. They rarely use a questionnaire mainly due to time constraints. According to the experience at the Sexual Rehabilitation Clinic of the University's General Hospital of Patras, 3 months is the usual time point when most patients come to the clinic after radical prostatectomy. In the first two months after surgery, patients are interested primarily in the oncological and continence issues and later they seek help for their erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Men above 18 years old wih clinically localized prostate cancer, who have undergone open or laparoscopic radical prostatectomy, with or without use of phosphoodiesterase-5 inhibitors

Exclusion Criteria:

* Penile anatomic defects
* Uncontrolled major medical illnesses such as uncontrolled diabetes, severe renal, hepatic or cardiovascular disease
* major psychiatrics disorders
* drug or alcohol abuse

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men above 18 years old wih clinically localized prostate cancer, who have undergone open or laparoscopic radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Score of recalled International Index of Erectile Function-5 | 3 months
  Score of recalled IIEF-5 collected 3 months after radical prostatectomy. The IIEF is a validated, brief and reliable self-administered questionnaire for assessing erectile function. The abridged five-item version of the 15-item IIEF possesses favorable properties for detecting the presence and severity of erectile dysfunction for the preceding 6 months. The IIEF-5 consists of five questions, each of which is scored on a five-point ordinal scale and erectile dysfunction may be classified into five categories based on the calculated scores. Based on IIEF-5 scores, erectile dysfunction severity is classified into the following five categories: severe (5±7), moderate (8±11), mild to moderate (12±16), mild (17±21), and no erectile dysfunction (22± 25).
Assessment of the degree of agreement between real time preoperative International Index of Erectile Function-5 score and recalled IIEF-5 3 months after radical prostatectomy | 3 months
  Assessment of the degree of agreement between real time preoperative IIEF-5 score and recalled IIEF-5 3 months after radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Kontogiannis, Study Director — University of Patras
Locations (1):
- University of Patras, Pátrai, Achaia, Greece